CLINICAL TRIAL: NCT06448975
Title: An Exploratory Study of Deep Cervical Lymphovenous Bypass (LVB) in Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19691027
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: Deep Cervical Lymphovenous Bypass; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The clinically diagnosed patients with mild to severe Alzheimer's Disease (Experimental): 1. The age ranged from 60 to 80 years, and the time from initial diagnosis to enrollment was more than 12 months
  2. The estimated survival time is more than 12 months;
  3. The clinically diagnosed patients with mild to severe Alzheimer's Disease;
  4. The imaging examination has the correlation diagnosis evidence;
  5. Volunteer to participate in the project and sign an informed consent form with the guardian.
  Interventions: Procedure: Deep cervical Lymphovenous Bypass

INTERVENTIONS:
Procedure: Deep cervical Lymphovenous Bypass — Deep cervical lymph-vein bypass surgery, connecting deep cervical lymph input vein vessel

SUMMARY:
The main pathological mechanism of Alzheimer's Disease (AD) is the abnormal deposition of amyloid-beta (Aβ) and tau proteins in the brain. Recent studies indicate that these two proteins are primarily cleared through the glymphatic system-meningeal lymphatic vessels-deep cervical lymphatic vessels pathway. Lymphatic circulation disorders in elderly patients can directly lead to the abnormal deposition of these proteins. Deep cervical lymphovenous bypass can improve lymphatic circulation and effectively treat lymphedema. This project aims to verify the effectiveness of 'deep cervical lymphovenous bypass' in treating AD, offering a new surgical treatment method to improve cognitive impairment and the quality of life for AD patients.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is a progressive neurodegenerative disorder that insidiously begins. Clinically characterized by memory impairment, aphasia, apraxia, agnosia, and other symptoms, it poses a severe threat to the quality of life of the elderly and brings a heavy burden to society and families. To date, there are no effective methods to prevent, halt, or cure AD. Therefore, there is an urgent need to explore new treatment approaches.

The definition of the glymphatic system and the discovery of meningeal lymphatic vessels (MLV) have overturned the traditional view of the immune privilege of the central nervous system, offering new clues and hope for the study and treatment of many brain diseases, including AD. The main pathological mechanism of Alzheimer's Disease (AD) is the abnormal deposition of amyloid-beta (Aβ) and tau proteins in the brain. Recent research indicates that these two proteins are primarily cleared through the glymphatic system-meningeal lymphatic vessels-deep cervical lymphatic vessels pathway, and lymphatic circulation disorders in elderly patients can directly lead to the abnormal deposition of these proteins. Deep cervical lymphovenous bypass can improve lymphatic circulation and effectively treat lymphedema. This project aims to verify the effectiveness of 'deep cervical lymphovenous bypass' in treating AD, providing a new surgical method to improve cognitive impairment and the quality of life for AD patients.

ELIGIBILITY:
Inclusion Criteria:

1. The age ranged from 60 to 80 years, and the time from initial diagnosis to enrollment was more than 12 months
2. The estimated survival time is more than 12 months;
3. The clinically diagnosed patients with mild to severe Alzheimer's Disease;
4. The imaging examination has the correlation diagnosis evidence;
5. Volunteer to participate in the project and sign an informed consent form with the guardian.

Exclusion Criteria:

1. Complicated with other severe systemic underlying diseases;
2. Unable to tolerate general anesthesia;
3. The pregnant women;
4. Recent severe infection or infectious diseases within 4 weeks;
5. Unable to complete the evaluator or refused to complete the one-year clinical follow-up.
6. Refusal to participate

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
PET scan | Baseline ,6 months ,12 months
  Detecting changes in the brain's amyloid and tau protein burden before and after surgery.Aβ/tau positron emission tomography (PET) facilitates spatial visualization and quantitative analysis of abnormal protein accumulations in the brains of Alzheimer's disease (AD) patients, offering objective imaging data crucial for early diagnosis, disease assessment, post-operative efficacy monitoring, and prognostic evaluations. Interpretations and quantitative assessments of Aβ-PET images are primarily focused on four cerebral regions: the lateral temporal cortex, frontal lobe, posterior cingulate gyrus/precuneus, and parietal lobe, aiding in the diagnosis of AD. The deposition of tau protein is positively correlated with disease severity; it initially accumulates predominantly in the medial temporal lobe and extends to neocortical regions during the middle and late stages. Tau PET is instrumental for monitoring disease progression and evaluating treatment outcomes.
The Alzheimer's Disease Comprehensive Rating Scale (iADRS) | Baseline ,1 week ,1 month ,3 months ,6 months ,12 months
  The change in iADRS scores before and after surgery. The iADRS is a simple linear combination of two recognized, treatment-sensitive, and widely accepted measures of Alzheimer's Disease (AD), namely the AD Assessment Scale-Cognitive Subscale (ADAS-Cog) and the Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-iADL), used for the measurement of core assessment domains in AD.The total score of ADAS-Cog ranges from 0 to 70, with higher scores indicating greater cognitive impairment. The total score of ADCS-iADL ranges from 0 to 78, assessing the ability to perform complex activities of daily living, with higher scores indicating greater functional impairment.

SECONDARY OUTCOMES:
Plasma Aβ1-42 and plasma p-tau181 | Baseline ,1 month ,6 months ,12 months
  Elevated preoperatively, postoperatively the indicators have decreased, with reference values being plasma Aβ1-42 ≤ 110.00 pg/mL; plasma p-tau181 ≤ 30.00 pg/mL.
Mini-Mental State Examination(MMSE) | Baseline ,1 week ,1 month ,3 months ,6 months ,12 months
  The MMSE score is a widely used brief cognitive assessment scale for the rapid screening of cognitive functions, especially dementia. It encompasses various aspects such as orientation to time, place, immediate memory, attention and calculation, delayed memory, language, and visuospatial abilities.The total score of MMSE is 0-30,with higher scores mean a better outcome.
Montreal Cognitive Assessment(MoCA) | Baseline ,1 week ,1 month ,3 months ,6 months ,12 months
  The MoCA (Montreal Cognitive Assessment) score is a specialized tool for the rapid screening of Mild Cognitive Impairment (MCI). The MoCA scale includes tests across various cognitive domains, such as attention and concentration, executive functions, memory, language, visuospatial skills, abstract thinking, calculation, and orientation, comprising a total of 11 examination items. The total score of the MoCA scale is 30 points, with a score of 26 points or above typically considered to indicate normal cognitive function, while a score below 26 may suggest the presence of cognitive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hua, Study Director — Affiliated Hosptial Of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China